CLINICAL TRIAL: NCT07022613
Title: The Impact of Mindfulness-Based Stress Reduction on Mindfulness, Self-Compassion, and Perceived Stress Among Healthcare Professionals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, birgül yazar, NURSE, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AkdenizU-SBF-BY-01
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Healthcare Professionals
Keywords: stress; Mindfulness; Self-Compassion; Healthcare Professionals; Occupational Health Nurse; Nursing
MeSH Terms: interventions — Perceived Stress Scale

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- program designed specifically for healthcare professionals, the intervention group (Experimental): In the first and last sessions, the Perceived Stress Scale (PSS), the Mindful Attention Awareness Scale (MAAS), the Self-Compassion Scale (SCS), and the Visual Analog Scale (VAS) will be administered, and saliva samples will be collected.
  In the remaining sessions, only the VAS-one of the stress measurement parameters-will be verbally administered. In this way, participants will be informed weekly about the progression of their stress levels.
  The program to be implemented in the study will consist of weekly sessions held over eight weeks. Each session will be conducted for groups of 10 participants, three consecutive days per week.
  Interventions: Other: Mindfulness-Based Stress Reduction Program
- control group (No Intervention): Participants will be interviewed twice: once at the beginning and once at the end of the intervention.During both the initial and final interviews, the Perceived Stress Scale (PSS), the Mindful Attention Awareness Scale (MAAS), the Self-Compassion Scale (SCS), and the Visual Analog Scale (VAS) will be administered, and saliva samples will be collected.

INTERVENTIONS:
Other: Mindfulness-Based Stress Reduction Program — The Mindfulness-Based Stress Reduction (MBSR) program is considered to offer healthcare professionals working under high levels of stress the opportunity to develop knowledge and skills in consciously recognizing their emotions, compassionately accepting painful feelings without suppression, and transforming negative thoughts and emotions into more constructive ones.
  In the first and last sessions, the Perceived Stress Scale (PSS), the Mindful Attention Awareness Scale (MAAS), the Self-Compassion Scale (SCS), and the Visual Analog Scale (VAS) will be administered, and saliva samples will be collected.
  In the remaining sessions, only the VAS-one of the stress measurement parameters-will be verbally administered. In this way, participants will be informed weekly about the progression of their stress levels.
  The program to be implemented in the study will consist of weekly sessions held over eight weeks. Each session will be conducted for groups of 10 participants, three consecutive days
  Other Names: Perceived Stress Scale; Mindful Attention Awareness Scale; A Scale to Mearsure Self-Compassion; Visual Analog Scale
  Arms: program designed specifically for healthcare professionals, the intervention group

SUMMARY:
Mindfulness is defined as a state of awareness in which an individual consciously pays attention to the present moment without judgment, reaction, or resistance, thereby promoting mental and psychological well-being.

Self-compassion refers to adopting a kind, understanding, and supportive attitude toward oneself. While mindfulness enables individuals to recognize sources of stress and develop strategies to cope with them, self-compassion encourages a gentle and caring approach toward oneself during this process. Research has shown that mindfulness practices enhance self-compassion and that these two constructs have a synergistic effect in reducing stress.

Work-related stress negatively affects both the professional functioning and overall health of individuals. Acknowledging the increasing prevalence of stress and stress-related illnesses, the International Labour Organization (ILO) officially included stress and stress-induced disorders in the list of occupational diseases in 2010. Compared to other professions, these stressors have a more profound physical and psychological impact on healthcare professionals. In this context, the concepts of mindfulness and self-compassion are critically important for enhancing the psychological resilience of healthcare professionals and improving their stress management skills.

This study is designed as a non-randomized, quasi-experimental pretest-posttest control group study to determine the effect of the Mindfulness-Based Stress Reduction (MBSR) program on the levels of mindfulness, self-compassion, and stress among healthcare professionals. Data collection tools will include a demographic information form, the Perceived Stress Scale (PSS), Mindful Attention Awareness Scale (MAAS), the A Scale to Mearsure Self-Compassion (SCS), and a Visual Analog Scale (VAS) for stress assessment. The research will be conducted with healthcare professionals working at Aksaray Training and Research Hospital, located in the central district of Aksaray, Turkey.

An 8-week Mindfulness-Based Stress Reduction (MBSR) program will be implemented for the intervention group. Data will be collected between May and December 2025. The results of the study will be analyzed using the Statistical Package for the Social Sciences (SPSS) version 25. In addition to standardized scales, the effectiveness of the MBSR program will also be evaluated using a biological stress marker-salivary cortisol.

The Mindfulness-Based Stress Reduction program implemented in this study is expected to contribute to the field of occupational health nursing. Furthermore, the program is anticipated to enhance healthcare professionals' abilities to consciously recognize their emotions, accept painful experiences with understanding rather than suppression, and transform negative thoughts and emotions into more constructive perspectives.

ELIGIBILITY:
Inclusion Criteria:

* The intervention group consisted of participants whose perceived stress levels were above the arithmetic mean, as measured by the Perceived Stress Scale
* Individuals who provided informed consent to participate in the study.

Exclusion Criteria:

* Individuals with communication impairments (e.g., hearing, vision, or speech difficulties)
* Individuals currently engaged in stress-reducing practices such as yoga or various forms of meditation
* Pregnant individuals
* Individuals receiving medical or psychosocial treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Participants will complete the scale once in the first phase of the study, and again during the first and final (eighth) weeks of the second phase."
  The Perceived Stress Scale (PSS) was developed by Cohen, Kamarck, and Mermelstein (1983).The PSS consists of 14 items and is designed to measure the degree to which situations in one's life are perceived as stressful. The internal consistency reliability of the scale, calculated based on item analysis, yielded a Cronbach's alpha coefficient of 0.84, and the test-retest correlation was found to be 0.87.
  Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very Often (4)." The scale comprises two subdimensions: perceived distress and perceived lack of control/self-efficacy. Items 1, 2, 3, 7, 11, 12, and 14 assess perceived distress, while items 4, 5, 6, 8, 9, 10, and 13 assess perceived lack of self-efficacy. Seven of the items, which are positively worded, are reverse scored. The total score on the PSS-14 ranges from 0 to 56, with higher scores indicating greater perceived stress.
Mindful Attention Awareness Scale | In the second phase of the study, the scale will be administered in both the first and the final (eighth) week.
  The Mindful Attention Awareness Scale (MAAS) was developed by Brown and Ryan (2003), and its Turkish validity and reliability study was conducted by Özyeşil et al. (2011).
  The scale has a Cronbach's alpha internal consistency coefficient of .80 and a test-retest correlation of .86. The MAAS measures the general tendency to be aware of and attentive to present-moment experiences in daily life.
  It consists of 15 items and is rated on a 6-point Likert-type scale (almost always, very frequently, sometimes, rarely, very rarely, almost never). The scale has a unidimensional structure and yields a single total score. Higher scores on the scale indicate higher levels of mindfulness.
A Scale to Mearsure Self-Compassion | In the second phase of the study, the scale will be administered in both the first and the final (eighth) week.
  The Self-Compassion Scale (SCS) was developed by Neff in 2003 and consists of 26 items.
  The scale measures six subdimensions: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. It is rated on a 5-point Likert-type scale (1 = Almost Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Almost Always).
  The overall reliability of the scale is high, with a Cronbach's alpha coefficient of .92. For the subscales, Cronbach's alpha values range between .75 and .81, indicating good internal consistency.
Visual Analog Scale | At the beginning of each session conducted with the intervention group in the second phase of the study, it is planned to use the Visual Analog Scale (VAS) to assess the participants' stress levels based on the previous week's evaluation.
  At the beginning of each session conducted with the intervention group in the second phase of the study, it is planned to use the Visual Analog Scale (VAS) to assess the participants' stress levels based on the previous week's evaluation.
  The Visual Analog Scale (VAS) is a tool used to convert subjective, non-quantifiable values into numerical data. It consists of a 10-centimeter horizontal line marked with numbers from 1 to 10 at one-centimeter intervals. The VAS is a well-established and widely accepted assessment instrument in the global scientific literature.Within the context of this study, a score of 10 on the Visual Analog Scale (VAS) will represent the highest level of perceived stress ('very stressed'), whereas a score of 0 will represent the absence of stress ('not stressed at all

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen E, Geiger P, Schiller C, Bluth K, Watkins L, Zhang Y, Xia K, Tauseef H, Leserman J, Girdler S, Gaylord S. Effects of Mindfulness-Based Stress Reduction on Experimental Pain Sensitivity and Cortisol Responses in Women With Early Life Abuse: A Randomized Controlled Trial. Psychosom Med. 2021 Jul-Aug 01;83(6):515-527. doi: 10.1097/PSY.0000000000000889. PMID 33259351